CLINICAL TRIAL: NCT05894798
Title: Acupuncture in Infantile Colic - A Randomised Trial.
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Region Skane (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 230524
Record Dates: First submitted 2023-05-24; First posted 2023-06-08 (Actual); Last update posted 2025-01-10 (Actual); Status verified 2024-10

CONDITIONS: Infant, Newborn, Diseases; Colic, Infantile; Acupuncture
Keywords: Infant colic; pain; primary healthcare; gastrointestinal
MeSH Terms: conditions — Infant, Newborn, Diseases; Colic; Pain | interventions — Acupuncture Therapy

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): The acupuncture nurse holds the child by the hand and speaks to it calmly for about a minute. The children receive acupuncture at point LI 4 in the grip of the thumb on the upper side of the hand, bilaterally, with a sterile disposable needle with dimensions 0.20 x 13 mm. The stitch is approximately three mm deep. The needle is allowed to remain in place for about 30 seconds
  Interventions: Other: Acupuncture
- Controll (No Intervention): The children in the control group do not receive acupuncture. However, they spend the same amount of time with the acupuncture nurse, are addressed and are touched in the same way as the children in the intervention group, but do not get stung.

INTERVENTIONS:
Other: Acupuncture — Acupuncture at point LI 4 in the thumb grip on the upper side of the hand, bilaterally, with a sterile disposable needle of dimension 0.20 x 13 mm. The stitch is approximately three mm deep. The needle is allowed to remain in place for about 30 seconds
  Arms: Intervention

SUMMARY:
About 10 per cent of all new born babies in Sweden have infant colic. This may affect the the whole family and the early connection between the baby and the parents. Although, there are no effective and safe treatment. Acupuncture is an environmental friendly method that affects pain, anxiety, sleep and the function of gastrointestinal system. Several studies have shown various results, and there are a need for high-qualitative randomised controlled trials to investigate the proposed effect further. 128 children will be randomised into two groups; acupuncture at LI4 or no acupuncture, parents will be blinded. Statistical calculations will be performed on the content of the diaries (bowel movement frequency, crying time, feeding). Registration of crying/crying in connection with acupuncture treatment, i.e. when the needle touches the skin or later until the needle is removed and 30 seconds after.

DETAILED DESCRIPTION:
Among all newborn babies in Sweden, about 10% have infant colic. Currently, there is no effective and safe treatment for infant colic, while there is an increase in the use of complementary methods to reduce the infant's suffering. Infant colic is defined as "crying and whining more than three hours/day more than three days/week" and affects about 10% of all newborn babies, starting when the baby is about two weeks old and usually stopping at 3-4 months of age. A complementary method used against pain in the Western world is acupuncture, a treatment method with ancient roots in Asia. It involves thin needles being inserted at specific points on the body. The needle sticks stimulate neurotransmitters, and hormones are released in the central nervous system. Acupuncture is an environmentally friendly treatment with few side effects and promotes the inherent ability to self-heal. Acupuncture has been shown in several studies to be a safe and effective method that affects pain, anxiety, sleep, and the function of the gastrointestinal system. Studies have shown both shorter crying time with lower intensity. Therefore, there is a reasonableness in acupuncture being able to alleviate infant colic. However, systematic reviews have not been able to show significant differences in symptoms between children who received acupuncture and those who did not. The reviews also described that the studies used different points on the body for treatment and that the acupuncture needles remained for various lengths of time (5-30 seconds). This led to their conclusion that more high-quality randomised studies are needed to investigate the treatment method further. Purpose To examine the effect of minimal acupuncture at a single point (LI4) on infants with colic compared to no acupuncture. Method: The parents register the baby's crying, feeding, sleep and bowel movements in a diary (appendix 1) for seven consecutive days, constituting a baseline. According to the diary registration, the infants who have colic are included and come twice a week for three weeks to a nurse at a selected child health centre (BVC). The children will be randomised into two groups; acupuncture at LI4 or no acupuncture. The parents will not know which group the child belongs to. The parents will fill in the same diary type as the baseline during the two intervention weeks. Statistical calculations will be performed on the content of the diaries (bowel movement frequency, crying time, feeding). Registration of crying/crying in connection with acupuncture treatment, i.e. when the needle touches the skin or later until the needle is removed and 30 seconds after. This registration will also be done in the control group, where the handling of children is the same but without acupuncture. Expected result This study can provide further evidence on whether acupuncture is an effective treatment method for alleviating symptoms of infant colic, as well as further highlighting any experience of pain associated with treatment. The attitude towards complementary approaches among parents with infants showing colic symptoms will also be investigated.

ELIGIBILITY:
Inclusion Criteria:

* Otherwise healthy infants, born in week 37 or later, aged 2 - 9 weeks who, according to diary entries, scream/whine for at least 3 hours/day for at least 3 days in the same week. The child has undergone a medical examination at BB or later with no pathological findings. The child takes no medicines or only the dietary supplement Semper Magdroppar. At least one parent understands and speaks Swedish.

Exclusion Criteria:

* Children who have lost more than one channel on their weight curve. Children who received acupuncture

Ages: 2 Weeks to 9 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 128 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Crying and screaming | During acupuncture
  Registration of crying and screaming during the acupuncture at each visit
Colic symptoms | Baseline to 3 weeks
  Change in colic symptoms during the treatment period, comparison between groups. information will be collected by the diaries the parents write during the intervention period

CONTACTS AND LOCATIONS:
Overall Officials: Veronica Milos Nymberg, Principal Investigator — Lund University/ Region Skane

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Savino F. Focus on infantile colic. Acta Paediatr. 2007 Sep;96(9):1259-64. doi: 10.1111/j.1651-2227.2007.00428.x. PMID 17718777
- [Background] Canivet C, Hagander B, Jakobsson I, Lanke J. Infantile colic--less common than previously estimated? Acta Paediatr. 1996 Apr;85(4):454-8. doi: 10.1111/j.1651-2227.1996.tb14060.x. PMID 8740304
- [Background] Talachian E, Bidari A, Rezaie MH. Incidence and risk factors for infantile colic in Iranian infants. World J Gastroenterol. 2008 Aug 7;14(29):4662-6. doi: 10.3748/wjg.14.4662. PMID 18698680
- [Background] Shamir R, St James-Roberts I, Di Lorenzo C, Burns AJ, Thapar N, Indrio F, Riezzo G, Raimondi F, Di Mauro A, Francavilla R, Leuchter RH, Darque A, Huppi PS, Heine RG, Bellaiche M, Levy M, Jung C, Alvarez M, Hovish K. Infant crying, colic, and gastrointestinal discomfort in early childhood: a review of the evidence and most plausible mechanisms. J Pediatr Gastroenterol Nutr. 2013 Dec;57 Suppl 1:S1-45. doi: 10.1097/MPG.0b013e3182a154ff. No abstract available. PMID 24356023
- [Background] Canivet C, Jakobsson I, Hagander B. Colicky infants according to maternal reports in telephone interviews and diaries: a large Scandinavian study. J Dev Behav Pediatr. 2002 Feb;23(1):1-8. doi: 10.1097/00004703-200202000-00001. PMID 11889345
- [Background] WESSEL MA, COBB JC, JACKSON EB, HARRIS GS Jr, DETWILER AC. Paroxysmal fussing in infancy, sometimes called colic. Pediatrics. 1954 Nov;14(5):421-35. No abstract available. PMID 13214956
- [Background] Landgren K, Hallstrom I. Parents' experience of living with a baby with infantile colic--a phenomenological hermeneutic study. Scand J Caring Sci. 2011 Jun;25(2):317-24. doi: 10.1111/j.1471-6712.2010.00829.x. Epub 2010 Aug 18. PMID 20723153
- [Background] Raiha H, Lehtonen L, Huhtala V, Saleva K, Korvenranta H. Excessively crying infant in the family: mother-infant, father-infant and mother-father interaction. Child Care Health Dev. 2002 Sep;28(5):419-29. doi: 10.1046/j.1365-2214.2002.00292.x. PMID 12296876
- [Background] Ellett ML, Appleton MM, Sloan RS. Out of the abyss of colic: a view through the fathers' eyes. MCN Am J Matern Child Nurs. 2009 May-Jun;34(3):164-71. doi: 10.1097/01.NMC.0000351704.35761.f1. PMID 19550259
- [Background] Landgren K, Lundqvist A, Hallstrom I. Remembering the Chaos - But Life Went on and the Wound Healed. A Four Year Follow Up with Parents having had a Baby with Infantile Colic. Open Nurs J. 2012;6:53-61. doi: 10.2174/1874434601206010053. Epub 2012 May 2. PMID 22655001
- [Background] Savino F, Tarasco V. New treatments for infant colic. Curr Opin Pediatr. 2010 Dec;22(6):791-7. doi: 10.1097/MOP.0b013e32833fac24. PMID 20859207
- [Background] Talvik I, Alexander RC, Talvik T. Shaken baby syndrome and a baby's cry. Acta Paediatr. 2008 Jun;97(6):782-5. doi: 10.1111/j.1651-2227.2008.00778.x. Epub 2008 Apr 7. PMID 18397351
- [Background] Myrhaug HT, Aas-Jakobsen E, Kjellemyr GT, Kirkehei I, Steen-Johnsen J, Havelsrud K, Helseth S. Treatment of Infant Colic [Internet]. Oslo, Norway: Knowledge Centre for the Health Services at The Norwegian Institute of Public Health (NIPH); 2009 Jun. Report from Norwegian Knowledge Centre for the Health Services (NOKC) No. 14-2009. Available from http://www.ncbi.nlm.nih.gov/books/NBK464835/ PMID 29320055
- [Background] Savino F, Pelle E, Palumeri E, Oggero R, Miniero R. Lactobacillus reuteri (American Type Culture Collection Strain 55730) versus simethicone in the treatment of infantile colic: a prospective randomized study. Pediatrics. 2007 Jan;119(1):e124-30. doi: 10.1542/peds.2006-1222. PMID 17200238
- [Background] Savino F, Cordisco L, Tarasco V, Palumeri E, Calabrese R, Oggero R, Roos S, Matteuzzi D. Lactobacillus reuteri DSM 17938 in infantile colic: a randomized, double-blind, placebo-controlled trial. Pediatrics. 2010 Sep;126(3):e526-33. doi: 10.1542/peds.2010-0433. Epub 2010 Aug 16. PMID 20713478
- [Background] Kukkonen K, Savilahti E, Haahtela T, Juntunen-Backman K, Korpela R, Poussa T, Tuure T, Kuitunen M. Long-term safety and impact on infection rates of postnatal probiotic and prebiotic (synbiotic) treatment: randomized, double-blind, placebo-controlled trial. Pediatrics. 2008 Jul;122(1):8-12. doi: 10.1542/peds.2007-1192. PMID 18595980
- [Background] Perry R, Hunt K, Ernst E. Nutritional supplements and other complementary medicines for infantile colic: a systematic review. Pediatrics. 2011 Apr;127(4):720-33. doi: 10.1542/peds.2010-2098. Epub 2011 Mar 28. PMID 21444591
- [Background] Posadzki P, Ernst E. Spinal manipulation: an update of a systematic review of systematic reviews. N Z Med J. 2011 Aug 12;124(1340):55-71. PMID 21952385
- [Background] Carlsson C. Acupuncture mechanisms for clinically relevant long-term effects--reconsideration and a hypothesis. Acupunct Med. 2002 Aug;20(2-3):82-99. doi: 10.1136/aim.20.2-3.82. PMID 12216606
- [Background] Macpherson H, Scullion A, Thomas KJ, Walters S. Patient reports of adverse events associated with acupuncture treatment: a prospective national survey. Qual Saf Health Care. 2004 Oct;13(5):349-55. doi: 10.1136/qhc.13.5.349. PMID 15465938
- [Background] Lin YC, Lee AC, Kemper KJ, Berde CB. Use of complementary and alternative medicine in pediatric pain management service: a survey. Pain Med. 2005 Nov-Dec;6(6):452-8. doi: 10.1111/j.1526-4637.2005.00071.x. PMID 16336482
- [Background] White A. A cumulative review of the range and incidence of significant adverse events associated with acupuncture. Acupunct Med. 2004 Sep;22(3):122-33. doi: 10.1136/aim.22.3.122. PMID 15551936
- [Background] Jindal V, Ge A, Mansky PJ. Safety and efficacy of acupuncture in children: a review of the evidence. J Pediatr Hematol Oncol. 2008 Jun;30(6):431-42. doi: 10.1097/MPH.0b013e318165b2cc. PMID 18525459
- [Background] Adams D, Cheng F, Jou H, Aung S, Yasui Y, Vohra S. The safety of pediatric acupuncture: a systematic review. Pediatrics. 2011 Dec;128(6):e1575-87. doi: 10.1542/peds.2011-1091. Epub 2011 Nov 21. PMID 22106073
- [Background] Gentry KR, McGinn KL, Kundu A, Lynn AM. Acupuncture therapy for infants: a preliminary report on reasons for consultation, feasibility, and tolerability. Paediatr Anaesth. 2012 Jul;22(7):690-5. doi: 10.1111/j.1460-9592.2011.03743.x. Epub 2011 Dec 6. PMID 22141917
- [Background] Kemper KJ, Sarah R, Silver-Highfield E, Xiarhos E, Barnes L, Berde C. On pins and needles? Pediatric pain patients' experience with acupuncture. Pediatrics. 2000 Apr;105(4 Pt 2):941-7. PMID 10742351
- [Background] Tsao JC, Zeltzer LK. Complementary and Alternative Medicine Approaches for Pediatric Pain: A Review of the State-of-the-science. Evid Based Complement Alternat Med. 2005 Jun;2(2):149-159. doi: 10.1093/ecam/neh092. Epub 2005 Apr 27. PMID 15937555
- [Background] Reinthal M, Lund I, Ullman D, Lundeberg T. Gastrointestinal symptoms of infantile colic and their change after light needling of acupuncture: a case series study of 913 infants. Chin Med. 2011 Aug 11;6:28. doi: 10.1186/1749-8546-6-28. PMID 21835014
- [Background] Baumler P, Zhang W, Stubinger T, Irnich D. Acupuncture-related adverse events: systematic review and meta-analyses of prospective clinical studies. BMJ Open. 2021 Sep 6;11(9):e045961. doi: 10.1136/bmjopen-2020-045961. PMID 34489268
- [Background] Ang L, Song E, Lee HW, Kim JT, Kim E, Lee MS. Acupuncture Treatment for Nocturnal Crying in Pediatric Patients: A Systematic Review of Clinical Studies. Front Pediatr. 2021 Jul 14;9:647098. doi: 10.3389/fped.2021.647098. eCollection 2021. PMID 34336731
- [Background] Zhao J. Treatment of infantile morbid night crying by acupuncture at Zhongchong point in 100 cases. J Tradit Chin Med. 2002 Mar;22(1):11. No abstract available. PMID 11977508
- [Background] Reinthal M, Andersson S, Gustafsson M, Plos K, Lund I, Lundeberg T, Gustaf Rosen K. Effects of minimal acupuncture in children with infantile colic - a prospective, quasi-randomised single blind controlled trial. Acupunct Med. 2008 Sep;26(3):171-82. doi: 10.1136/aim.26.3.171. PMID 18818563
- [Background] Landgren K, Kvorning N, Hallstrom I. Acupuncture reduces crying in infants with infantile colic: a randomised, controlled, blind clinical study. Acupunct Med. 2010 Dec;28(4):174-9. doi: 10.1136/aim.2010.002394. Epub 2010 Oct 18. PMID 20959312
- [Background] Landgren K, Kvorning N, Hallstrom I. Feeding, stooling and sleeping patterns in infants with colic--a randomized controlled trial of minimal acupuncture. BMC Complement Altern Med. 2011 Oct 11;11:93. doi: 10.1186/1472-6882-11-93. PMID 21989212
- [Background] Landgren K, Hallstrom I. Effect of minimal acupuncture for infantile colic: a multicentre, three-armed, single-blind, randomised controlled trial (ACU-COL). Acupunct Med. 2017 Jun;35(3):171-179. doi: 10.1136/acupmed-2016-011208. Epub 2017 Jan 16. PMID 28093383
- [Background] Skjeie H, Skonnord T, Fetveit A, Brekke M. Acupuncture for infantile colic: a blinding-validated, randomized controlled multicentre trial in general practice. Scand J Prim Health Care. 2013 Dec;31(4):190-6. doi: 10.3109/02813432.2013.862915. Epub 2013 Nov 15. PMID 24228748
- [Background] Skjeie H, Skonnord T, Fetveit A, Brekke M. A pilot study of ST36 acupuncture for infantile colic. Acupunct Med. 2011 Jun;29(2):103-7. doi: 10.1136/aim.2010.003590. Epub 2011 Mar 29. PMID 21450707
- [Background] Lee D, Lee H, Kim J, Kim T, Sung S, Leem J, Kim TH. Acupuncture for Infantile Colic: A Systematic Review of Randomised Controlled Trials. Evid Based Complement Alternat Med. 2018 Oct 24;2018:7526234. doi: 10.1155/2018/7526234. eCollection 2018. PMID 30473718
- [Background] Skjeie H, Skonnord T, Brekke M, Klovning A, Fetveit A, Landgren K, Hallstrom IK, Brurberg KG. Acupuncture treatments for infantile colic: a systematic review and individual patient data meta-analysis of blinding test validated randomised controlled trials. Scand J Prim Health Care. 2018 Mar;36(1):56-69. doi: 10.1080/02813432.2018.1426146. Epub 2018 Jan 17. PMID 29338487
- See also: SBU - Swedish Agency for Health Technology Assessment and Assessment of Social Services. Does acupuncture relieve colic? (in Swedish) — https://www.sbu.se/contentassets/861e18c230c347e082a7e9be256a29f1/sbu_ut_lindras_kolik_av_akupunktur.pdf
- See also: Rikshandboken i barnhälsovård (in Swedish; The national handbook in child health care) — https://www.rikshandboken-bhv.se/pediatrik/buk---oversikt/spadbarnskolik/